CLINICAL TRIAL: NCT05390203
Title: Sexual Function Before and After Bariatric Surgeries.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Abdelrheem Abouelfotouh Abdulrahaman Kenawy Elbakh, Andrology Specialist, Assiut University
Other Study IDs: ED and Bariatric surgeries
Record Dates: First submitted 2022-05-06; First posted 2022-05-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Sexual Dysfunction
MeSH Terms: conditions — Sexual Dysfunction, Physiological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Penile duplex study, Hormonal Assay (Total Testosterone, Prolactin and E2) — we will do penile duplex and hormonal profile preoperatively and 6 months postoperatively.

SUMMARY:
To assess sexual function before and the impact of weight loss after bariatric surgery among obese men with sexual dysfunction.

DETAILED DESCRIPTION:
Obesity is a worldwide prevalent problem which is currently considered a pandemic disease. It is intimately related to several comorbidities that negatively impact physical and mental health. Male sexual dysfunction is not uncommon in people with obesity. This could be attributed to many obesity-associated conditions as diabetes mellitus (DM), hypertension (HTN), and mental and social impairment. Obesity indirectly affects male sexual function by inducing many comorbidities associated with sexual dysfunction. Obesity is also a complex endocrine disorder that can independently alter sexual function through the disruption of various sex hormones. Men with morbid obesity often suffer from deep but reversible sexual dysfunction. Several managements have been introduced to deal with obesity. Dietary intervention, medications, physical exercise are widely used in case of mild and moderate obesity. Meanwhile, bariatric surgery has become the most effective treatment strategy for morbid obese patients which can bring great weight reduction and is expected to ameliorate the comorbidities. Mora et al.'s prospective study showed a bariatric surgery-related significant increase in the IIEF score at 1 year postoperatively. This was found also by the Groutz et al. and Kun et al. However, in a retrospective study by Rosenblatt et al., there was no significant increase in the IIEF scores following RYGB surgery in 23 male patients. Similarly, Sarwer et al., in their prospective study, found that despite the increased postoperative IIEF scores, this difference lied out of significance except for the overall satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* The study will involve fifty-five obese male patients "those indicated for bariatric surgery" complaining from sexual dysfunction with score ≤ 21 in the International Index of Erectile Function-5 (IIEF-5) questionnaire.

N.B. Indication for bariatric surgeries when they have BMI ≥ 40 kg/m2 or ≥ 35 kg/m2 with comorbidities.

Exclusion Criteria:

* Patients who are not married;
* Those with severe psychic illness.
* And those with congenital or acquired penile problems interfere with sexual intercourse.

Ages: 18 Years to 60 Years | Sex: Male
Age Groups: Adult
Gender Based: Yes
Study Population: The study will involve fifty-five obese male patients "those indicated for bariatric surgery" complaining from sexual dysfunction with score ≤ 21 in the International Index of Erectile Function-5 (IIEF-5) questionnaire.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Assessing Sexual function before and after bariatric surgeries. | We will assess the scores of the questionnaire preoperatively and the change of each score at 6 months postoperatively to evaluate if there are changes after bariatric surgery on sexual function or not.
  Assessing Sexual function (Erectile function, Orgasmic function, sexual desire, intercourse satisfaction and overall satisfaction) after bariatric surgery by the International Index of Erectile Function (IIEF)-5 questionnaire preoperatively and 6 months postoperatively.
  International Index of Erectile Function-IIEF-5) as a diagnostic tool for ED. The possible scores for the IIEF-5 range from 5 to 25, and ED was classified into five categories based on the scores: severe (5-7), moderate (8-11), mild to moderate (12-16), mild (17-21), and no ED (22-25)

SECONDARY OUTCOMES:
Penile Duplex Doppler Data, Hormonal Profile Data and patients' demographic data. | Will be assessed preoperatively and 6 months postoperatively.
  we will assess Weight by kilogram, Height by centimeter and BMI by Kg/m2. Our patients are candidate for bariatric surgeries when they have BMI ≥ 40 kg/m2 or ≥ 35 kg/m2 with comorbidities.
  Normal values for Total testesterone is from 1.6 to 7.8 ng/ml. Normal values for Prolactin is less than 20 ng/ml. Normal values for Estradiol (E2) is up to 39.8 pg/ml.

CONTACTS AND LOCATIONS:
Overall Officials: EmadEldin Kamal Ali, PHD, Study Director — Professor of Andrology , Assiut University; Osama Yassin Mostafa Taha, Principal Investigator — Professor of plastic surgery, Assiut University; Ahmed Mahmoud Mohamed Abdellah, Study Chair — Lecturer of Andrology , Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Meldrum DR, Morris MA, Gambone JC. Obesity pandemic: causes, consequences, and solutions-but do we have the will? Fertil Steril. 2017 Apr;107(4):833-839. doi: 10.1016/j.fertnstert.2017.02.104. Epub 2017 Mar 11. PMID 28292617
- [Background] Djalalinia S, Qorbani M, Peykari N, Kelishadi R. Health impacts of Obesity. Pak J Med Sci. 2015 Jan-Feb;31(1):239-42. doi: 10.12669/pjms.311.7033. PMID 25878654
- [Background] Esfahani SB, Pal S. Obesity, mental health, and sexual dysfunction: A critical review. Health Psychol Open. 2018 Jul 12;5(2):2055102918786867. doi: 10.1177/2055102918786867. eCollection 2018 Jul-Dec. PMID 30023076
- [Background] Di Vincenzo A, Busetto L, Vettor R, Rossato M. Obesity, Male Reproductive Function and Bariatric Surgery. Front Endocrinol (Lausanne). 2018 Dec 18;9:769. doi: 10.3389/fendo.2018.00769. eCollection 2018. PMID 30619096
- [Background] Dallal RM, Chernoff A, O'Leary MP, Smith JA, Braverman JD, Quebbemann BB. Sexual dysfunction is common in the morbidly obese male and improves after gastric bypass surgery. J Am Coll Surg. 2008 Dec;207(6):859-64. doi: 10.1016/j.jamcollsurg.2008.08.006. Epub 2008 Oct 1. PMID 19183532
- [Background] Efthymiou V, Hyphantis T, Karaivazoglou K, Gourzis P, Alexandrides TK, Kalfarentzos F, Assimakopoulos K. The effect of bariatric surgery on patient HRQOL and sexual health during a 1-year postoperative period. Obes Surg. 2015 Feb;25(2):310-8. doi: 10.1007/s11695-014-1384-x. PMID 25085222
- [Background] Colquitt JL, Pickett K, Loveman E, Frampton GK. Surgery for weight loss in adults. Cochrane Database Syst Rev. 2014 Aug 8;2014(8):CD003641. doi: 10.1002/14651858.CD003641.pub4. PMID 25105982
- [Background] Picot J, Jones J, Colquitt JL, Gospodarevskaya E, Loveman E, Baxter L, Clegg AJ. The clinical effectiveness and cost-effectiveness of bariatric (weight loss) surgery for obesity: a systematic review and economic evaluation. Health Technol Assess. 2009 Sep;13(41):1-190, 215-357, iii-iv. doi: 10.3310/hta13410. PMID 19726018
- [Background] Mora M, Aranda GB, de Hollanda A, Flores L, Puig-Domingo M, Vidal J. Weight loss is a major contributor to improved sexual function after bariatric surgery. Surg Endosc. 2013 Sep;27(9):3197-204. doi: 10.1007/s00464-013-2890-y. Epub 2013 Apr 24. PMID 23612762
- [Background] Groutz A, Gordon D, Schachter P, Amir H, Shimonov M. Effects of bariatric surgery on male lower urinary tract symptoms and sexual function. Neurourol Urodyn. 2017 Mar;36(3):636-639. doi: 10.1002/nau.22980. Epub 2016 Feb 16. PMID 26879634
- [Background] Kun L, Pin Z, Jianzhong D, Xiaodong H, Haoyong Y, Yuqian B, Hongwei Z. Significant improvement of erectile function after Roux-en-Y gastric bypass surgery in obese Chinese men with erectile dysfunction. Obes Surg. 2015 May;25(5):838-44. doi: 10.1007/s11695-014-1465-x. PMID 25361762